CLINICAL TRIAL: NCT01914770
Title: Effectiveness of Belimumab Treatment in a Subpopulation of Systemic Lupus Erythematosus (SLE) Patients: a Pooled Analysis of BLISS-52 and BLISS-76
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 114246
Record Dates: First submitted 2012-04-03; First posted 2013-08-02 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2013-09

CONDITIONS: Systemic Lupus Erythematosus
Keywords: pooled analyses; quality of life; SELENA SLEDAI; SLE; steroid use; responder rate; flares; belimumab; BILAG
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with systemic lupus erythematosus (SLE): Subjects with SLE receiving ongoing stable SLE treatment
  Interventions: Drug: Belimumab 1 mg/kg; Drug: Belimumab 10 mg/kg; Drug: Placebo

INTERVENTIONS:
Drug: Belimumab 1 mg/kg — Subjects received belimumab 1 mg/kg in addition to their ongoing stable systemic lupus erythematosus (SLE) treatment regimen. Belimumab was administered intravenously at 0, 2, 4 weeks and every 4 weeks thereafter. The ongoing SLE treatment regimen was to have been stable for at least 30 days prior to Day 0, which consisted of any of the following (alone or in combination): prednisone or equivalent (from 0 to 40 mg/day when used in combination with other SLE treatment or from 7.5 to 40 mg/day alone), anti-malarials, non-steroidal anti inflammatory drugs (NSAIDs), or any immunosuppressive therapy (ie, methotrexate, azathioprine, leflunomide, or mycophenolate calcineurin inhibitors, sirolimus, oral cyclophosphamide, 6-mercaptopurine, or thalidomide).
Drug: Belimumab 10 mg/kg — Subjects received belimumab 10 mg/kg in addition to their ongoing stable SLE treatment regimen. Belimumab was administered intravenously at 0, 2, 4 weeks and every 4 weeks thereafter. The ongoing SLE treatment regimen was to have been stable for at least 30 days prior to Day 0, which consisted of any of the following (alone or in combination): prednisone or equivalent (from 0 to 40 mg/day when used in combination with other SLE treatment or from 7.5 to 40 mg/day alone), anti-malarials, NSAIDs, or any immunosuppressive therapy (ie, methotrexate, azathioprine, leflunomide, or mycophenolate calcineurin inhibitors, sirolimus, oral cyclophosphamide, 6-mercaptopurine, or thalidomide).
Drug: Placebo — Subjects received placebo in addition to their ongoing stable SLE treatment regimen. Placebo was administered intravenously at 0, 2, 4 weeks and every 4 weeks thereafter. The ongoing SLE treatment regimen was to have been stable for at least 30 days prior to Day 0, which consisted of any of the following (alone or in combination): prednisone or equivalent (from 0 to 40 mg/day when used in combination with other SLE treatment or from 7.5 to 40 mg/day alone), anti-malarials, NSAIDs, or any immunosuppressive therapy (ie, methotrexate, azathioprine, leflunomide, or mycophenolate calcineurin inhibitors, sirolimus, oral cyclophosphamide, 6-mercaptopurine, or thalidomide).

SUMMARY:
This pooled analysis will assess data from the Phase 3 belimumab registration studies BLISS-52 (aka BEL110752) and BLISS-76 (aka BEL110751). The analysis was pre-planned and agreed prior to the unblinding of either study. The primary objective is to evaluate the impact of belimumab treatment on a more severe subpopulation of systemic lupus erythematosus (SLE) subjects from BLISS-52 and BLISS-76 to aid physicians and payers in decision making. Subjects are from the modified Intent-to-Treat (ITT) population defined as randomized subjects who received at least 1 dose of study agent. This more severe subpopulation will have renal, neurological, haematological, or cardiovascular/respiratory organ domain involvement (as defined by a British Isles Lupus Assessment Group (BILAG) domain score of A, B or C in at least one of the domains) at baseline AND anti-double-stranded deoxyribonucleic acid (anti-dsDNA) positive (≥ 30 IU/mL) at baseline OR low C3 and/or C4 complement relative to the normal range at baseline.

ELIGIBILITY:
Inclusion Criteria

* Eligible subjects for BLISS-52 and BLISS-76 included:
* clinical diagnosis of systemic lupus erythematosus (SLE) according to the American College of Rheumatology (ACR) criteria
* "active" (systemic lupus erythematosus) SLE disease, defined as a safety of oestrogen in lupus national assessment (SELENA) systemic lupus erythematosus disease activity index (SLEDAI) disease activity score of at least 6 at screening
* an unequivocally positive antinuclear antibodies (ANA) test result, from 2 independent time points within the study screening period or 1 positive historical test result and 1 positive test result during the screening period. ANA test results obtained in the screening period were only considered positive if the ANA titer ≥ 1:80 and/or anti-dsDNA serum antibody was ≥ 30 IU/mL
* on a stable SLE treatment regimen for at least 30 days prior to Day 0, which consisted of any of the following (alone or in combination): prednisone or equivalent (from 0 to 40 mg/day when used in combination with other SLE treatment or from 7.5 to 40 mg/day alone), anti-malarials, non-steroidal anti inflammatory drugs (NSAIDs), or any immunosuppressive therapy (i.e., methotrexate, azathioprine, leflunomide, or mycophenolate calcineurin inhibitors, sirolimus, oral cyclophosphamide, 6-mercaptopurine, or thalidomide).
* Additional inclusion criteria for the purpose of this analysis: subpopulation of patients from the pooled modified Intent-to-Treat population from BLISS-52 and BLISS-76 who have renal, neurological, haematological, or cardiovascular/respiratory organ domain involvement (as defined by a BILAG domain score of A, B or C in at least one of the domains) at baseline and 1 of the following:

  * are anti-dsDNA positive (≥ 30 IU/mL) at baseline, OR
  * have low C3 and/or C4 complement relative to the normal range at baseline.

Exclusion Criteria:

* Key exclusion criteria for BLISS-52 and BLISS-76 included:
* severe active lupus nephritis or Central Nervous System (CNS) lupus
* pregnancy
* receipt of any B cell target therapy at any time
* receipt of an investigational agent within 60 days prior to Day 0 for non-biologics and within 1 year for biologics
* receipt of abatacept (within 1 year), intravenous (IV) cyclophosphamide (within 6 months), anti-tumor necrosis factor (anti-TNF) therapy, anakinra, IV immunoglobulin (IVIG), prednisone > 100 mg/day, or plasmapheresis within 3 months, or live vaccine within 1 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary population is the subpopulation of patients from the pooled modified Intent-to-Treat population from BLISS-52 and BLISS-76 who have renal, neurological, haematological, or cardiovascular/respiratory organ domain involvement (as defined by a BILAG domain score of A, B or C in at least one of the domains) at baseline and 1 of the following:
  * are anti-double-stranded deoxyribonucleic acid (anti-dsDNA) positive (= 30 IU/mL) at baseline, OR
  * have low C3 and/or C4 complement relative to the normal range at baseline.
Sampling Method: Probability Sample
Enrollment: 1016 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Responder Rate | Week 52
  Response is defined as: ≥4 point reduction from baseline in SELENA SLEDAI score, no worsening (increase of < 0.30 points from baseline) in PGA, and no new BILAG A organ domain score or 2 new BILAG B organ domain scores.

SECONDARY OUTCOMES:
SELENA SLEDAI | Week 52
  Percent of subjects with ≥ 4 point reduction from baseline in SELENA SLEDAI score at Week 52
SF-36 | Week 24
  Mean change in SF-36 Health Survey physical component summary score (PCS) at Week 24
Time to first flare by SLE Flare Index | Up to Week 52
  Time to 1st SLE flare after 24 weeks by modified SLE Flare Index

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline